CLINICAL TRIAL: NCT03100084
Title: The PREPPeD Study: "PREdelivery Placental Biomarkers- Pregnancy and Delivery Outcome"
Brief Title: PREdelivery Placental Biomarkers- Pregnancy and Delivery Outcome
Acronym: PREPPeD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian SIDS and Stillbirth Society (Other); Extrastiftelsen (Other)
Responsible Party: Principal Investigator, Meryam Sugulle, Consultant Obstetrician, Oslo University Hospital
Other Study IDs: 36864; 36259 (Other: Oslo University Hospital)
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Pregnancy Complications; Placental Insufficiency
Keywords: Preeclampsia; Diabetes in Pregnancy; Fetal Growth Restriction; Reduced Fetal Movements
MeSH Terms: conditions — Pregnancy Complications; Placental Insufficiency; Pre-Eclampsia; Diabetes, Gestational; Fetal Growth Retardation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal plasma, serum and DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- I. Post Dates: Pregnant women referred for clinical post term evaluation and/or labour induction.
  Blood sampling.
  Interventions: Other: Blood sampling
- II. Induction of Labour: Pregnant women ≥37+0 GW (gestational week) referred for labour induction (any cause).
  Blood sampling.
  Interventions: Other: Blood sampling
- III. All Outpatients: Pregnant women ≥37+0 GW presenting for any medical reason at OUH outpatient clinic.
  Blood sampling
  Interventions: Other: Blood sampling
- IV. Diabetes in Pregnancy: Pregnant women ≥36+0 GW with pregestational or gestational diabetes. Blood sampling.
  Interventions: Other: Blood sampling
- V. Reduced Fetal Movements: Pregnant women ≥37+0 GW with reduced fetal movements and/or referred due to reduced symphysis-fundal height.
  Blood sampling.
  Interventions: Other: Blood sampling
- VI. Hypertensive Disorders in Pregnancy: Pregnant women referred for preeclampsia (or other pregnancy induced hypertensive disorders) and/or suspected fetal growth restriction; longitudinal cohorts.
  Blood sampling.
  Interventions: Other: Blood sampling
- VII. All Labour Admissions: All pregnant women ≥37+0 GW admitted for labour. Blood sampling.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Maternal blood sampling

SUMMARY:
The PREPPeD study proposes that predelivery placenta-derived maternal circulating biomarkers reflect placental health, capacity and ageing, and can help predict onset and complications of delivery both in complicated pregnancies as well as in clinically uncomplicated term/post-term pregnancies.

DETAILED DESCRIPTION:
The main aim of the PREPPeD study is to explore whether placental health, evaluated by maternal blood biomarkers in late pregnancy, correlates with delivery outcomes in both healthy and complicated pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women scheduled to deliver at the Department of Obstetrics at OUH who qualify for the study groups as specified in the "Groups and Intervention" section.

Exclusion Criteria:

* Women who do not understand Norwegian or English
* Communicable disease
* Younger than 18 years of age
* Legally incompetent
* Fetal malformations

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: All pregnant women scheduled to deliver at the Department of Obstetrics at OUH who qualify for the study groups as specified in the "Groups and Intervention" section.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-09-15 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Fetal acidaemia | Umbilical cord gas/lactate are sampled directly post partum within 45 min; data assessed throughout study period of 140 months
  In neonates delivered by cesarean section (CS) without labour (defined as absence of regular uterine contractions):
  Umbilical artery blood (transporting blood from the fetus to the placenta) pH<7.13 and arterial BD >10.0
  In neonates from labored delivery (regardless of subsequent delivery method, vaginal or CS):
  Umbilical artery blood pH<7.05 and arterial BD>14; OR Umbilical artery blood (or venous if arterial blood not available) lactate above Reference level for respective gestational age according to publication by Wiberg N et al ,BJOG 2008 (doi: 10.1111/j.1471-0528.2008.01707.x.)
Newborn low Apgar score | Apgar score is assessed directly post partum within 10 minutes; data assessed throughout study period of 140 months
  <4 at 1 minute OR <7 at 5 minutes
Newborn asphyxia | Directly post partum within 10 and 45 minutes respectively; data assessed throughout study period of 140 months
  Combination of outcomes 1 and 2
Rate of intrauterine fetal demise/intra-/postpartum fetal death | Diagnosis within 28 days postpartum; data assessed throughout study period of 140 months
Neonatal intubation/mechanical ventilation>6 hours | Within 28 days postpartum; data assessed throughout study period of 140 months
Meconium aspiration syndrome | Diagnosis within 28 days postpartum; data assessed throughout study period of 140 months
Neonatal hypoxic-ischemic encephalopathy | Diagnosis within 28 days postpartum; data assessed throughout study period of 140 months
Therapeutic hypothermia of the neonate | Within 3 days postpartum; data assessed throughout study period of 140 months
Rate of acute cesarean section (due to suspected fetal distress) | Data assessed throughout study period of 140 months

SECONDARY OUTCOMES:
Rates of operative vaginal deliveries (forceps/vacuum/combined; due to suspected fetal distress) | Data assessed throughout study period of 140 months
Pathological placenta histology findings | Data assessed throughout study period of 140 months
Abnormal intrapartum CTG patterns | Intrapartum CTG; data assessed throughout study period of 140 months

CONTACTS AND LOCATIONS:
Overall Officials: Meryam Sugulle, PhD, MD, Principal Investigator — Oslo University Hospital, Department of Obstetrics
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Depending on when the permission for the dataset usage for the project's outcome measures ends (OUH personal data officer/Regional Ethical Comittee) AND Norwegian legislation regarding personal data protection. It is unlikely that a major part of the data set will be shared openly due to these restrictions on sensitive personal data matters.

REFERENCES:
- [Derived] Mitlid-Mork B, Turowski G, Bowe S, Staff AC, Sugulle M. Circulating angiogenic profiles and histo-morphological placental characteristics of uncomplicated post-date pregnancies. Placenta. 2021 Jun;109:55-63. doi: 10.1016/j.placenta.2021.04.017. Epub 2021 May 5. PMID 33990027